CLINICAL TRIAL: NCT00289991
Title: Prospective, Open-Label, Comparative, Multi-Center Study Of Voriconazole Compared To Itraconazole For The Primary Prophylaxis Of Invasive Fungal Infection (IFI) With Allogeneic Hematopoietic Stem Cell Transplants (HSCT)
Brief Title: Voriconazole Versus Itraconazole In Primary Prophylaxis Of Invasive Fungal Infection (IFI) In Subjects With Allogeneic Hematopoietic Stem Cell Transplants (HSCT)
Acronym: IMPROVIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A1501073
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Antifungal Prophylaxis of Invasive Fungal Infections
MeSH Terms: interventions — Itraconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itraconazole (Active Comparator)
  Interventions: Drug: Itraconazole
- Voriconazole (Experimental)
  Interventions: Drug: Vfend - voriconazole

INTERVENTIONS:
Drug: Itraconazole — Prophylaxis
  Arms: Itraconazole
Drug: Vfend - voriconazole — Prophylaxis
  Other Names: Vfend
  Arms: Voriconazole

SUMMARY:
Study is to compare antifungal prophylaxis of Voriconazole and Itraconazole in subjects who have had a Stem Cell Transplant. The success of the end point will be measured using evidence of Infection, drug compliance and survival.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT for acute leukemia (AML, ALL or myelodysplastic syndrome) failed lymphoma therapy or transformation of CML
* Male and Female over 12 years or greater

Exclusion Criteria:

* Possible, probable or proven IFI at study entry or at any time in 6 months prior to study entry, defined according to the 'consensus criteria' (Ascioglu et al 2002)
* Previous history of zygomycosis
* Anticipated survival less than one month

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2006-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- Canada (4):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Bmo
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Cairo, Egypt
- France (8):
  - Pfizer Investigational Site, Marseille, Cedex 09
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Villejuif
- Greece (2):
  - Pfizer Investigational Site, Exohi Asvestohoriou, Thessaloniki
  - Pfizer Investigational Site, Athens
- Pfizer Investigational Site, Amman, Jordan
- Portugal (2):
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Spain (6):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Salamanca, Salamanca
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Switzerland (2):
  - Pfizer Investigational Site, Ch-4031 Basel
  - Pfizer Investigational Site, Geneva
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Kayseri
- United Kingdom (9):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501073

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were stratified at the time of randomization by the following factors: conditioning regimen (myeloablative or non-myeloablative); relatedness of donor (matched/related or mismatched/unrelated).
Groups:
- Voriconazole: Voriconazole (tablet or powder for oral suspension) loading dose regimen intravenous (IV) for first 24 hours: 6 milligrams per kilogram (mg/kg) of body weight every 12 hours; maintenance dose (after first 24 hours) 4 mg/kg of body weight (IV) twice daily (BID) or 200 mg tablet or powder for oral suspension by mouth (PO) BID (subjects greater than or equal to [≥] 40 kg body weight) or 100 mg tablet or powder for oral suspension twice daily (subjects less than [<] 40 kg body weight).
- Itraconazole: Itraconazole (Sporanox™ Liquid) oral solution 200 mg PO BID. Loading dose as IV formulation on Days 0 and 1.
Period: Overall Study
Arm/Group | Voriconazole | Itraconazole
Started | 234 | 255
Completed | 176 | 175
Not Completed | 58 | 80
Not completed — Death | 35 | 38
Not completed — Adverse Event | 15 | 13
Not completed — Failure of prophylaxis | 1 | 1
Not completed — Fungal breakthrough infection | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 12
Not completed — Other | 5 | 14

BASELINE CHARACTERISTICS:
Groups:
- Voriconazole: Voriconazole (tablet or powder for oral suspension) loading dose regimen IV for first 24 hours: 6 mg/kg of body weight every 12 hours; maintenance dose (after first 24 hours) 4 mg/kg of body weight (IV) BID or 200 mg tablet or powder for oral suspension PO BID (subjects ≥ 40 kg body weight) or 100 mg tablet or powder for oral suspension twice daily (subjects < 40 kg body weight).
- Total: Total of all reporting groups
Arm/Group | Voriconazole | Itraconazole | Total
Number analyzed (Participants) | 234 | 255 | 489
Age, Customized [Number; unit: participants]
  <18 years | 9 | 11 | 20
  Between 18 and 44 years | 106 | 119 | 225
  Between 45 and 64 years | 104 | 115 | 219
  >=65 years | 15 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.4) | 42.7 (14.6) | 43.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 100 | 196
  Male | 138 | 155 | 293

OUTCOME MEASURES:

1. Primary Outcome: Success at Day 180: Percent of Responders (Randomization Strata)
Description: Percent of responders (by randomization strata) with success of antifungal prophylaxis at 180 days after allogeneic hematopoietic stem cell transplant (HSCT). Success: alive at Day 180 (Visit 9), had not developed a breakthrough proven or probable invasive fungal infection (IFI) by Visit 9, and received full course of study drug prophylaxis without interruption of greater than 14 days in total during the prophylaxis period; defined as failure if these criteria were not met. Additionally, if subject withdrew from study completely before Visit 9, imputed as failure at Visit 9 (programmatically).
Time Frame: Day 180 (Visit 9)
Population: Modified Intent to Treat (MITT): primary analysis population; all randomized subjects: received at least 1 dose of randomized study drug and had allogeneic HSCT; data from 1 site excluded due to Good Clinical Practice (GCP) deviations; (n)=number of subjects with analyzable data at observation for voriconazole and itraconazole, respectively.
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants
  Myeloablative/matched related (n=66, 85) | 59.1 | 44.7
  Myeloablative/mismatched unrelated (n=59, 58) | 52.5 | 25.9
  Non-myeloablative/matched related (n=58, 57) | 34.5 | 28.1
  Non-myeloablative/mismatched unrelated (n=41, 41) | 46.3 | 26.8
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Non-inferiority inferred if lower limit of the 2-sided 95 percent (%) confidence interval (CI) for the difference between the voriconazole and itraconazole treatment groups in the adjusted proportion of subjects classified as "Success" at Day 180 after transplant is above -10%. Superiority achieved if 2-sided 95% CI for difference between these treatment groups in the adjusted proportion of subjects classified as "Success" at Day 180 after transplant does not include zero and is positive; Test type: Non-Inferiority or Equivalence — Assuming a true success rate of 50% in voriconazole (Vori) treatment (Tx) group and 45% in itraconazole (Itra) Tx group, sample size of 232 subjects per group=90% power to demonstrate non-inferiority of Vori to Itra using pre-specified non-inferiority margin of -10%. Sample has at least 80% power to demonstrate superiority of Vori over Itra if true success rates for Vori and Itra are 57% and 44% respectively. Based on this, up to 500 subjects were to be enrolled to obtain 464 eligible subjects; Difference in adjusted responder rates; Difference in adjusted responder rates using Fleiss method; percent difference adjusted proportions = 16.4, 95% CI 2-sided [7.7 to 25.1] — Overall treatment difference in adjusted proportions (expressed as percentages) calculated using Fleiss method

2. Secondary Outcome: Success at Day 100: Percent of Responders (Randomization Strata)
Description: Percent of responders (by randomization strata) with success of antifungal prophylaxis at 100 days after allogeneic HSCT. Success defined as: alive at Day 100 (Visit 7), had not developed a breakthrough proven or probable IFI by Visit 7, and received full course of study drug prophylaxis without an interruption of >14 days in total during the prophylaxis period; defined as failure if these criteria were not met. Additionally, if subject withdrew from study completely before Visit 7, imputed as failure at Visit 7 (programmatically).
Time Frame: Day 100 (Visit 7)
Population: MITT; data from 1 site excluded due to GCP deviations; (n)=number of subjects with analyzable data at observation for voriconazole and itraconazole, respectively.
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants
  Myeloablative/matched related (n=66, 85) | 65.2 | 50.6
  Myeloablative/mismatched unrelated (n=59, 58) | 55.9 | 27.6
  Non-myeloablative/matched related (n=58, 57) | 43.1 | 38.6
  Non-myeloablative/mismatched unrelated (n=41, 41) | 48.8 | 36.6
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Test type: Non-Inferiority or Equivalence — Non-inferiority inferred if lower limit of the 2-sided 95% confidence interval (CI) for the difference between the voriconazole and itraconazole treatment groups in the adjusted proportion of subjects classified as "Success" at Day 100 after transplant is above -10%. Superiority achieved if 2-sided 95% CI for difference between these treatment groups in the adjusted proportion of subjects classified as "Success" at Day 100 after transplant does not include zero and is positive; Difference in adjusted responder rates; Difference in adjusted responder rates using the Fleiss method; percent difference adjusted proportions = 15.4, 95% CI 2-sided [6.6 to 24.2] — Overall treatment difference in adjusted proportions (expressed as percentages) calculated using Fleiss method

3. Secondary Outcome: Time to Breakthrough Invasive Fungal Infection (IFI)
Description: Summary of time (in days) from start of prophylaxis to first recorded occurrence of breakthrough proven or probable IFI.
Time Frame: Day 1 up to Day 180 (Visit 9)
Population: MITT; data from 1 site excluded due to GCP deviations. Analysis excludes additional data on IFIs that were only captured on European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) worksheets (not on Case Report Forms or in the database). Times were summarized only for subjects who experienced a breakthrough IFI.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 3 | 4
days | 119.0 (28.58) [48.0 to 190.0] | 77.0 (77.08) [0.0 to 199.6]

4. Secondary Outcome: Percent of Subjects With Occurrence of Breakthrough IFI
Description: Percent of subjects with occurrence of breakthrough IFI (proven or probable). Included all subjects in the MITT population.
Time Frame: Day 1 up to Day 100 (Visit 7) and Day 180 (Visit 9)
Population: MITT; data from 1 site excluded due to GCP deviations. Analysis excludes additional data on IFIs that were only captured on EORTC/MSG worksheets (not on Case Report Forms or in the database).
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants
  Day 100 | 0.9 | 1.2
  Day 180 | 1.3 | 1.7
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Day 100; difference in proportions (expressed as percentages), voriconazole relative to itraconazole; Test type: Superiority or Other; p = 0.7114, Difference in proportions; Difference in proportions (approximate result); difference in proportions: percent = -0.4, 95% CI 2-sided [-2.2 to 1.5] — Approximate 2-sided 95 percent (%) confidence interval for the difference in proportions
Statistical Analysis 2: Comparison: Voriconazole vs Itraconazole; Day 180; difference in proportions (expressed as percentages), voriconazole relative to itraconazole; Test type: Superiority or Other; p = 0.7759, Difference in proportions; Difference in proportions (approximate result); difference in proportion: percent = -0.3, 95% CI 2-sided [-2.5 to 1.9] — Approximate 2-sided 95 percent (%) confidence interval for the difference in proportions

5. Secondary Outcome: Survival: Percent of Subjects Who Died at or Before Day 180
Description: Percent of subjects who died at or before Day 180, derived from the crude death rate. All subjects in the MITT population included in this proportion.
Time Frame: Day 1 up to Day 180 (Visit 9)
Population: MITT; data from 1 site excluded due to GCP deviations. Analysis does not include any deaths recorded in the long-term follow-up data (not available at time of analysis).
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants | 15.6 | 15.4
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Day 180; difference in proportions (expressed as a percentage), voriconazole relative to itraconazole; Test type: Superiority or Other; Difference in proportions; Difference in proportions (approximate result); difference in proportions: percent = 0.3, 95% CI 2-sided [-6.3 to 6.9] — Approximate 2-sided 95% confidence interval for the difference in proportions

6. Secondary Outcome: Time to Discontinuation of Study Treatment
Description: Time in days to discontinuation of study treatment defined as the number of days from first dose to last dose inclusive as recorded in the dosing log.
Time Frame: Day 1 up to Day 180 (Visit 9)
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
days | 88.7 (61.41) [80.6 to 96.8] | 71.5 (52.21) [64.9 to 78.2]
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Mann-Whitney test used to investigate the null hypothesis that the times to discontinuation of study medication in each treatment group come from the same distribution; Test type: Superiority or Other; p = 0.0026, Wilcoxon (Mann-Whitney); 2-sided Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Survival: Percent of Subjects Who Died Within 1 Year
Description: Percent of subjects who died within 1 year after transplant, derived from the crude death rate. All subjects in the MITT population included in this proportion. Only deaths up until and including 365 days after first dose of study medication included in the analysis.
Time Frame: Day 1 up to 1 year (Day 365)
Population: MITT; data from 1 site excluded due to GCP deviations. Typically, subjects received first dose study treatment on the day of their transplant; however, some subjects started treatment up to 48 hours after transplant. Data summarized with first day of study medication defined as Day 1.
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants | 25.9 | 30.7
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Day 365; difference in proportions (expressed as a percentage), voriconazole relative to itraconazole; Test type: Superiority or Other; p = 0.2487, Difference in proportions; Difference in proportions (approximate result); difference in proportions: percent = -4.8, 95% CI 2-sided [-13.0 to 3.4] — Approximate 2-sided 95 percent % confidence interval for the difference in proportions

8. Secondary Outcome: Duration of Treatment
Description: Median duration in days of treatment. Treatment is defined as the total number of days on which subjects took medication.
Time Frame: Day 1 up to Day 180
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Median (Full Range); unit: days
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
days | 96.0 [1 to 258] | 68.0 [3 to 223]

9. Secondary Outcome: Percent of Subjects With Use of Other Systemic Antifungal Agents as Empirical or Therapeutic Treatment
Description: Percent of subjects who used other systemic antifungal agents as empirical or therapeutic treatment, defined as either empirical: subject took a systemic antifungal agent at any time after the day of first dose of medication and did not develop a breakthrough proven or probable IFI during the study or therapeutic: subject developed a breakthrough proven or probable IFI.
Time Frame: Day 1 up to Day 180
Population: MITT; data from 1 site excluded due to GCP deviations. Subjects who developed a breakthrough proven or probable IFI were identified only from the study database, not the EORTC/MSG worksheet. In addition, all agents identified to be antifungals were considered to be systemic.
Measure: Number; unit: percent of participants
Arm/Group | Voriconazole | Itraconazole
Number analyzed (Participants) | 224 | 241
percent of participants | 40.6 | 49.4
Statistical Analysis 1: Comparison: Voriconazole vs Itraconazole; Difference in proportions (expressed as a percentage), voriconazole relative to itraconazole; Test type: Superiority or Other; p = 0.0570, Difference in proportions; Difference in proportions (approximate result); difference in proportions: percent = -8.8, 95% CI 2-sided [-17.8 to 0.3] — Approximate 2-sided 95% confidence interval for the difference in proportions

ADVERSE EVENTS:
Arm/Group | Voriconazole | Itraconazole
Serious Adverse Events (participants affected / at risk) | 111/234 | 95/255
Other Adverse Events (participants affected / at risk) | 228/234 | 252/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=234) | Itraconazole (N=255)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Disbacteriosis (Gastrointestinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 6
Retching (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 7
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 19 | 11
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 3 | 3
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 1
Acute graft versus host disease (Immune system disorders) | 2 | 7
Acute graft versus host disease in intestine (Immune system disorders) | 5 | 6
Acute graft versus host disease in liver (Immune system disorders) | 5 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0
Bone marrow transplant rejection (Immune system disorders) | 1 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 3
Graft versus host disease (Immune system disorders) | 9 | 8
Transplant rejection (Immune system disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 2
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 2
Central line infection (Infections and infestations) | 3 | 0
Ear infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 4 | 4
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 4
Septic shock (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 9 | 11
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 1 | 1
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung injury (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 4 | 0
Cytomegalovirus antigen positive (Investigations) | 0 | 1
Cytomegalovirus test (Investigations) | 2 | 2
Cytomegalovirus test positive (Investigations) | 2 | 1
Gram stain positive (Investigations) | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Weight (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Disseminated large cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 3 | 6
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Subdural haematoma evacuation (Surgical and medical procedures) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=234) | Itraconazole (N=255)
Anaemia (Blood and lymphatic system disorders) | 30 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 35 | 41
Febrile neutropenia (Blood and lymphatic system disorders) | 51 | 68
Neutropenia (Blood and lymphatic system disorders) | 21 | 30
Tachycardia (Cardiac disorders) | 13 | 6
Visual impairment (Eye disorders) | 15 | 2
Constipation (Gastrointestinal disorders) | 41 | 21
Diarrhoea (Gastrointestinal disorders) | 100 | 132
Abdominal discomfort (Gastrointestinal disorders) | 12 | 5
Abdominal pain (Gastrointestinal disorders) | 45 | 50
Abdominal pain upper (Gastrointestinal disorders) | 23 | 21
Dyspepsia (Gastrointestinal disorders) | 25 | 22
Nausea (Gastrointestinal disorders) | 86 | 91
Vomiting (Gastrointestinal disorders) | 78 | 103
Haemorrhoids (Gastrointestinal disorders) | 12 | 10
Oral pain (Gastrointestinal disorders) | 15 | 12
Stomatitis (Gastrointestinal disorders) | 17 | 17
Catheter related complication (General disorders) | 11 | 13
Catheter site erythema (General disorders) | 16 | 10
Pyrexia (General disorders) | 105 | 101
Asthenia (General disorders) | 19 | 31
Chest pain (General disorders) | 13 | 11
Chills (General disorders) | 17 | 23
Fatigue (General disorders) | 35 | 19
Mucosal inflammation (General disorders) | 115 | 142
Oedema (General disorders) | 13 | 13
Oedema peripheral (General disorders) | 37 | 42
Cholestasis (Hepatobiliary disorders) | 14 | 10
Cytolytic hepatitis (Hepatobiliary disorders) | 15 | 8
Hepatotoxicity (Hepatobiliary disorders) | 19 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 13
Acute graft versus host disease (Immune system disorders) | 12 | 16
Graft versus host disease (Immune system disorders) | 36 | 36
Folliculitis (Infections and infestations) | 12 | 11
Upper respiratory tract infection (Infections and infestations) | 12 | 8
Cytomegalovirus infection (Infections and infestations) | 22 | 17
Haemoglobin decreased (Investigations) | 13 | 8
Alanine aminotransferase increased (Investigations) | 12 | 4
Liver function test abnormal (Investigations) | 17 | 9
Weight increased (Investigations) | 10 | 13
Anorexia (Metabolism and nutrition disorders) | 19 | 25
Decreased appetite (Metabolism and nutrition disorders) | 9 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 | 30
Fluid overload (Metabolism and nutrition disorders) | 4 | 17
Fluid retention (Metabolism and nutrition disorders) | 14 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 30
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 24
Headache (Nervous system disorders) | 63 | 69
Tremor (Nervous system disorders) | 11 | 19
Dizziness (Nervous system disorders) | 13 | 9
Paraesthesia (Nervous system disorders) | 14 | 5
Anxiety (Psychiatric disorders) | 15 | 18
Insomnia (Psychiatric disorders) | 23 | 17
Renal failure (Renal and urinary disorders) | 19 | 12
Dysuria (Renal and urinary disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 22
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 12
Erythema (Skin and subcutaneous tissue disorders) | 43 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 24
Rash (Skin and subcutaneous tissue disorders) | 48 | 45
Petechiae (Skin and subcutaneous tissue disorders) | 7 | 13
Hypotension (Vascular disorders) | 16 | 18
Hypertension (Vascular disorders) | 44 | 49

LIMITATIONS AND CAVEATS:
Data was excluded from 1 site due to Good Clinical Practices deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.